CLINICAL TRIAL: NCT00002678
Title: Comparative Study of Dexamethasone vs Prednisone (Both in Combination With Melphalan) as Induction Therapy in Untreated Symptomatic Myeloma With an Additional Assessment of Dexamethasone vs no Additional Treatment as Maintenance Therapy in Non-Progressing Patients
Brief Title: Combination Chemotherapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY7; CAN-NCIC-MY7 (Other: PDQ); NCI-V95-0713 (Other: NCI); CDR0000064328 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melphan plus prednisone (Active Comparator): melphalan plus prednisone qd x 4 28 day cycles x 12 cycles; No treatment after stable response.
  Interventions: Drug: melphalan; Drug: prednisone
- Melphan, prednisone pluse dexamethasone (Active Comparator): melphalan plus prednisone qd x 4 28 day cycles x 12 cycles; dexamethasone qd x 4 q 28 days after non-progression
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 40 mg daily for four days given orally and repeated every 28 days should commence on day 29 of the twelfth cycle of induction therapy.
  Arms: Melphan, prednisone pluse dexamethasone
Drug: melphalan — 9 mg/m2 daily for 4 days given orally on an empty stomach every 4 weeks
  Arms: Melphan plus prednisone
Drug: prednisone — 100 mg daily for 4 days given orally on a full stomach with each cycle of melphalan
  Arms: Melphan plus prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective in treating patients with multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of various combination chemotherapy regimens in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with previously untreated stage I-III multiple myelome treated with melphalan combined with dexamethasone or prednisone as induction therapy.
* Compare the overall survival of patients with stable or responding disease after induction treated with dexamethasone vs observation alone as maintenance therapy.
* Compare the time to progression, response rate, and quality of life of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, stage (I or II vs III), creatinine (less than 2.0 mg/dL vs 2.0 mg/dL or greater), and intention to use prophylactic bisphosphonate (yes vs no).

* Induction: Patients are randomized to 1 of 4 treatment arms.

  * Arms I and II: Patients receive induction comprising oral prednisone followed by oral melphalan on days 1-4.
  * Arms III and IV: Patients receive induction comprising oral melphalan and oral dexamethasone (DM) on days 1-4 of all courses and DM on days 15-18 of courses 1-3.

Induction for arms I-IV continues every 4 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after induction proceed to maintenance therapy.

* Maintenance:

  * Arms I and III: Patients undergo observation.
  * Arms II and IV: Patients receive oral DM on days 1-4. Maintenance therapy continues every 4 weeks for arms II and IV and every 3 months for arms I and III in the absence of disease progression or unacceptable toxicity. Patients on arms I-IV who develop disease progression proceed to reinduction.
* Reinduction: Patients restart induction on the arm to which they were originally randomized. Reinduction continues every 4 weeks in the absence of stable response lasting 16 weeks, disease progression, or unacceptable toxicity. Patients who achieve a stable response lasting 16 weeks restart maintenance therapy. Patients who experience further disease progression during reinduction are taken off study.

Quality of life is assessed at baseline, on day 1 of courses 1-3 and then every 3 courses during induction, and then every 3 months during maintenance therapy.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A maximum of 600 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven previously untreated stage I-III multiple myeloma

  * Patients with stage I disease must be symptomatic
* Must meet at least 1 of the following conditions:

  * Plasma cells in osteolytic lesion or soft tissue tumor biopsy
  * At least 10% plasmacytosis in bone marrow aspirate and/or biopsy
  * Less than 10% plasma cells in bone marrow but at least 1 bony lesion
* Detectable serum M-component of IgG, IgA, IgD, or IgE

  * If only light chain disease (urine M-protein) present, urinary excretion of light chain (Bence Jones) protein must be at least 1.0 g/24 hours

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-4

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent serious illness
* Concurrent diabetes allowed, at the discretion of the treating physician, if changes in insulin requirements can be managed
* No other prior or concurrent malignancy except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunizations
* No concurrent filgrastim (G-CSF) or other growth factors as prophylaxis
* Concurrent epoetin alfa for anemia allowed

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior dexamethasone or prednisone with radiotherapy for spinal cord compression allowed if cumulative dexamethasone dose no greater than 120 mg and cumulative prednisone dose no greater than 792 mg
* Prior or concurrent corticosteroids for hypercalcemia allowed

Radiotherapy:

* See Endocrine therapy
* Prior focal radiotherapy allowed
* Concurrent focal radiotherapy during induction allowed
* Concurrent radiotherapy for palliation (e.g., painful osteolytic lesions or spinal cord compression) allowed

Surgery:

* At least 2 years since prior surgery for radiologic or endoscopic diagnosis of gastric or duodenal ulcer

Other:

* At least 2 years since prior medication for radiologic or endoscopic diagnosis of gastric or duodenal ulcer
* Prior or concurrent bisphosphonates for hypercalcemia allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 1995-06-02 (Actual); Primary Completion 2004-05-03 (Actual); Study Completion 2009-12-21 (Actual)

PRIMARY OUTCOMES:
Overall survival | 9 years
  To compare overall survival between:
  i) patients receiving melphalan-prednisone and those receiving melphalan-dexamethasone as induction therapy ii) patients maintained by dexamethasone and those on no additional treatment in the subgroup whose disease has not progressed at the time of the 12th induction cycle

SECONDARY OUTCOMES:
Time to progression | 9 years
Response rates | 9 years
Toxicity | 9 years
Quality of Life | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Shustik, MD, Study Chair — Royal Victoria Hospital - Montreal
Locations (37):
- St. Mary's/Duluth Clinic Health System, Duluth, Minnesota, United States
- Canada (36):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Providence Health Care - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - McGill University, Montreal, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shustik C, Belch A, Robinson S, Rubin SH, Dolan SP, Kovacs MJ, Grewal KS, Walde D, Barr R, Wilson J, Gill K, Vickars L, Rudinskas L, Sicheri DA, Wilson K, Djurfeldt M, Shepherd LE, Ding K, Meyer RM. A randomised comparison of melphalan with prednisone or dexamethasone as induction therapy and dexamethasone or observation as maintenance therapy in multiple myeloma: NCIC CTG MY.7. Br J Haematol. 2007 Jan;136(2):203-11. doi: 10.1111/j.1365-2141.2006.06405.x. PMID 17233817
- [Result] Shustik C, Belch A, Robinson S, et al.: Dexamethasone (dex) maintenance versus observation (obs) in patients with previously untreated multiple myeloma: a National Cancer Institute of Canada Clinical Trials Group study: MY.7. [Abstract] J Clin Oncol 22 (Suppl 14): A-6510, 560s, 2004.
- [Result] Shustik C, Belch A, Meyer R, et al.: Melphalan-dexamethasone is not superior to melphalan-prednisone as induction therapy in multiple myeloma. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1191, 2001.